CLINICAL TRIAL: NCT05657236
Title: Effect of Strength and Conditioning Training on Functional Performance in Children With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chronic kidney disease
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Diseases; plyometric exercises; muscle strength; balance
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other)
  Interventions: Other: medical treatment
- Experimental group (Experimental)
  Interventions: Other: medical treatment; Other: plyometric exercise

INTERVENTIONS:
Other: medical treatment — traditional medical treatment and regular follow-up
Other: plyometric exercise — Each session starts with a 5-minute warm-up of flexibility exercises (active range motion and stretching exercises).The main plyometric exercise set will be applied for 20-30 minutes and consisted of 10 exercises directed at the lower body that gradually progress by increasing the set/repetition number in two exercise blocks, each continue for 1 month .The cool down period is 5 minutes and includes walking at self-preferred speed and static stretches of the major muscle groups.
  Arms: Experimental group

SUMMARY:
Despite the benefits of physical rehabilitation among adults and children with chronic illness, they avoid to engage in different physical activities especially pediatric population. Most of the children with Chronic kidney disease receive their medical treatment and follow-up with no change of their functional performance. We still lack the evidence of plyometric exercises in pediatric population with Chronic kidney disease . Therefore, the primary aim of this study is to explore the effects of strength and conditioning training in the form of plyometric exercises on balance and muscle strength in children with Chronic kidney disease .

ELIGIBILITY:
Inclusion Criteria:

* Age will be ranged from 6-10 years.
* Both genders were included.
* Can follow instructions.
* Medically stable sedentary children with CKD, GFR (stage 2 (mild) eGFR of 60-89 ml/min per 1.73 m2, stage 3 (moderate) eGFR 30-59 ml/min per 1.73 m2) stage 4 (severe) eGFR of 15-29 ml/min per 1.73 m2.
* Did not yet require renal replacement therapy (non-dialysis).

Exclusion Criteria:

* Recent myocardial infarction, uncontrolled hypertension, unstable angina, symptomatic left ventricular fibrillation.
* Severe uncontrolled diabetes,
* Neurological or cognitive disorders
* Peripheral vascular disease.

Ages: 6 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Balance | after 2 months
  The Human Assessment Computer (HUMAC), a computerized dynamic posturography (commuter sports medicine, Inc., Stoughton, MA),will be used in the current study.
muscle strength | after 2 months
  The Laffayette manual muscle testing (model 01163 USA) is used for objectively quantifying muscle strength including hip flexors and abductors; knee flexors and extensors

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Mahmoud, Principal Investigator — Cairo university, faculty of physical therapy; Amira M Al-tohamy, Study Chair — Cairo university, faculty of physical therapy; Rasha M Helmy, Study Director — Cairo University
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt